CLINICAL TRIAL: NCT06398301
Title: The Effect of Surgical Prehabilitation on Autonomic Nervous System Regulation
Brief Title: Surgical Prehabilitation on Autonomic Nervous System (TUNE)
Acronym: TUNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Giulia Veronesi (Unknown); Katia Donadello (Unknown)
Responsible Party: Principal Investigator, Giovanni Landoni, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TUNE - CET 199-2023
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Surgery
Keywords: Thoracic surgery; Prehabilitation; Multimodal prehabilitation program; Standard care treatment; Hospital stay; Functional walking; Nutrition; Diet; Exercise; Relaxation; Functional recovery; Anesthesiology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Prehabilitation arm groups will receive preoperative intervention which includes exercise training, nutritional therapy and anxiety reducing techniques, aimed at preventing or attenuating surgery-driven functional decline.
  Interventions: Behavioral: Multimodal prehabilitation Program
- Control group (No Intervention): Standard care treatment. Application of ERAS pathways (Enhanced Recovery After Surgery)

INTERVENTIONS:
Behavioral: Multimodal prehabilitation Program — A tailored intervention will be prescribed if specific physical, nutritional or psychological impairments will be identified during the assessment phase. Based on the data obtained during the multimodal assessment, different domains and levels of care will be prescribed, focusing on exercise training, and/or nutrition optimization, and/or distress-coping techniques. Different combinations of three domains will be utilized to maximize their synergistic anabolic effect.
  The duration of program will be set at 4 weeks. All activities will be performed in dedicated suites at each site, under supervision of qualified health professionals.
  Arms: Prehabilitation

SUMMARY:
This study will be a multicenter interventional randomized trial evaluating the effect of a multimodal prehabilitation program on heart rate variability (HRV). In the same protocol the impact of HRV on hospital length of stay will be identified. One hundred patients aged 18 years or older scheduled for elective surgery will be eligible for enrolment, if they will not present any exclusion criteria. Patients will be randomized with a 1:1 allocation to receive either prehabilitation or standard of care.

DETAILED DESCRIPTION:
There is a growing interest whether prehabilitation interventions can reduce length of hospital stay and perioperative morbidity after major surgery. The aim of prehabilitation is to improve patients' functional capacity to withstand the upcoming stress of surgery. Prehabilitation is defined as an active program of structured exercise over a period of weeks to improve preoperative cardiovascular, respiratory, and muscular conditioning. Exercise in preparation for surgery is known to be associated with reduced postoperative complications and rapid restoration of functional status. However, prehabilitation programs are not yet standardized and there is no consensus on which parameters can accurately evaluate their effectiveness.

Many elements of prehabilitation are analogous to athletes' training, and it seems straightforward to compare prehabilitation before surgery to athletic preparation before competitions. Traditionally, post training recovery and physiological reserve are assessed by tools considered expensive and challenging in everyday use. For this reason, the use of heart rate variability (HRV), the variability in the distance between the R-R waves of the electrocardiogram, has become a logical solution as it identifies major regulatory processes after exercise. HRV parameters are commonly used to analyze stress experienced by the body during training and they can predict physiological recovery after training. HRV is the most validated method to measure the activity of the sympathetic and parasympathetic nervous systems. Surgery is considered as a physical stress which the body responds to by means of sympathetic and parasympathetic nervous system activities. While on one hand the sympathetic nervous system upregulates mechanisms of body response in stress situations, parasympathetic system is activated during relaxation through the vagus nerve. Among the effects of the sympathetic nervous system there are hyperglycemia, increased blood pressure and heart rate, activation of the inflammatory response, and increased myocardial oxygen consumption. Sympathetic nervous system activity tends to synchronize with the R-R intervals, reducing their variability. HRV measures the balance between parasympathetic and sympathetic nervous systems, and it seems to be associated to perioperative hypotension, nociception/anesthesia balance, and perioperative risk assessment. The reduction in the risk of coronary artery disease following physical activity may be due to increased HRV. Similarly, surgical prehabilitation could have beneficial effects on perioperative outcome through a possible increase in HRV.

Therefore, the aim of this study is to evaluate the impact of a multimodal program of prehabilitation on heart rate variability in patients undergoing thoracic surgery. Patients enrolled in this study will be randomized (ratio 1:1) and allocated either to the intervention group (Prehabilitation), or to the control group, which will be treated according to usual standard of care within Enhanced Recovery After Surgery (ERAS) pathways. The hypothesis is that standard deviation of normal to normal index of heart rate variability from baseline to the days before surgery will increase in patients undergoing prehabilitation. The hypothesis is also to observe a reduction of length of hospital stays in patient with an elevated standard deviation of normal to normal index of heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo major thoracic surgery including lobectomy, bilobectomy, anatomical segmentectomy, and pneumonectomy with general anesthesia;
* Patients ≥18 years of age at the time of randomization;
* Patients who provide written informed consent to participate.

Exclusion Criteria:

* New York Heart Association classes 3-4;
* End-stage organ dysfunction;
* American Society of Anesthesiologists physical status classes 4-5;
* Disabling orthopedic, neuromuscular, and psychiatric diseases;
* Other medical conditions that preclude safe training.
* Atrial fibrillation or other arrhythmia (e.g. bigeminy, trigeminy) that preclude heart rate variability analysis.
* Unable to provide written informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Impact of prehabilitation on heart rate variability | 30 days after prehabilitation
  The primary outcome measure will be standard deviation of normal to normal index (SDNN) of heart rate variability from baseline to the days before surgery.

SECONDARY OUTCOMES:
Lenght of hospital stay | 60 days follow up post surgery
  Reduction of length of hospital stay

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS San Raffaele Scientific Institute, Milan
  - Università degli studi di Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinstein AS, Sigurdsson MI, Bader AM. Comparison of Preoperative Assessment of Patient's Metabolic Equivalents (METs) Estimated from History versus Measured by Exercise Cardiac Stress Testing. Anesthesiol Res Pract. 2018 Sep 3;2018:5912726. doi: 10.1155/2018/5912726. eCollection 2018. PMID 30250484
- [Background] Pedziwiatr M, Mavrikis J, Witowski J, Adamos A, Major P, Nowakowski M, Budzynski A. Current status of enhanced recovery after surgery (ERAS) protocol in gastrointestinal surgery. Med Oncol. 2018 May 9;35(6):95. doi: 10.1007/s12032-018-1153-0. PMID 29744679
- [Background] Pedziwiatr M, Kisialeuski M, Wierdak M, Stanek M, Natkaniec M, Matlok M, Major P, Malczak P, Budzynski A. Early implementation of Enhanced Recovery After Surgery (ERAS(R)) protocol - Compliance improves outcomes: A prospective cohort study. Int J Surg. 2015 Sep;21:75-81. doi: 10.1016/j.ijsu.2015.06.087. Epub 2015 Jul 29. PMID 26231994
- [Background] Scheede-Bergdahl C, Minnella EM, Carli F. Multi-modal prehabilitation: addressing the why, when, what, how, who and where next? Anaesthesia. 2019 Jan;74 Suppl 1:20-26. doi: 10.1111/anae.14505. PMID 30604416
- [Background] Carli F, Zavorsky GS. Optimizing functional exercise capacity in the elderly surgical population. Curr Opin Clin Nutr Metab Care. 2005 Jan;8(1):23-32. doi: 10.1097/00075197-200501000-00005. PMID 15585997
- [Background] Wynter-Blyth V, Moorthy K. Prehabilitation: preparing patients for surgery. BMJ. 2017 Aug 8;358:j3702. doi: 10.1136/bmj.j3702. No abstract available. PMID 28790033
- [Background] Orange ST, Northgraves MJ, Marshall P, Madden LA, Vince RV. Exercise prehabilitation in elective intra-cavity surgery: A role within the ERAS pathway? A narrative review. Int J Surg. 2018 Aug;56:328-333. doi: 10.1016/j.ijsu.2018.04.054. Epub 2018 May 3. PMID 29730070
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Manou-Stathopoulou V, Korbonits M, Ackland GL. Redefining the perioperative stress response: a narrative review. Br J Anaesth. 2019 Nov;123(5):570-583. doi: 10.1016/j.bja.2019.08.011. Epub 2019 Sep 20. PMID 31547969
- [Background] McCorry LK. Physiology of the autonomic nervous system. Am J Pharm Educ. 2007 Aug 15;71(4):78. doi: 10.5688/aj710478. PMID 17786266
- [Background] Anderson TA. Heart rate variability: implications for perioperative anesthesia care. Curr Opin Anaesthesiol. 2017 Dec;30(6):691-697. doi: 10.1097/ACO.0000000000000530. PMID 28957877
- [Background] Paris A, Tonner PH, Bein B, von Knobelsdorff G, Scholz J. [Heart rate variability in anesthesia]. Anaesthesiol Reanim. 2001;26(3):60-9. German. PMID 11455865
- [Background] Aubert AE, Seps B, Beckers F. Heart rate variability in athletes. Sports Med. 2003;33(12):889-919. doi: 10.2165/00007256-200333120-00003. PMID 12974657
- [Background] Bernardi L, Valle F, Coco M, Calciati A, Sleight P. Physical activity influences heart rate variability and very-low-frequency components in Holter electrocardiograms. Cardiovasc Res. 1996 Aug;32(2):234-7. doi: 10.1016/0008-6363(96)00081-8. PMID 8796109
- [Background] Nunan D, Sandercock GR, Brodie DA. A quantitative systematic review of normal values for short-term heart rate variability in healthy adults. Pacing Clin Electrophysiol. 2010 Nov;33(11):1407-17. doi: 10.1111/j.1540-8159.2010.02841.x. PMID 20663071
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Carli F, Gillis C, Scheede-Bergdahl C. Promoting a culture of prehabilitation for the surgical cancer patient. Acta Oncol. 2017 Feb;56(2):128-133. doi: 10.1080/0284186X.2016.1266081. Epub 2017 Jan 9. PMID 28067101
- [Background] Colado JC, Pedrosa FM, Juesas A, Gargallo P, Carrasco JJ, Flandez J, Chupel MU, Teixeira AM, Naclerio F. Concurrent validation of the OMNI-Resistance Exercise Scale of perceived exertion with elastic bands in the elderly. Exp Gerontol. 2018 Mar;103:11-16. doi: 10.1016/j.exger.2017.12.009. Epub 2017 Dec 17. PMID 29262307